CLINICAL TRIAL: NCT03033329
Title: A Randomized, Double-Blind, Placebo Controlled Three-Part Study of the Safety, Tolerability, and Pharmacokinetics of MRX 4 Administered Intravenously to Healthy Volunteers in Single Ascending and Multiple Ascending Dose Cohorts, and Bioavailability of Oral MRX-4 Versus Intravenous Administration
Brief Title: Single Dose Escalation and Multiple Dose Escalation Trial of an Intravenous Formulation of MRX-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicuRx (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRX4-002
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2017-01

CONDITIONS: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Single intravenous doses of MRX-4 (Experimental): Single escalating intravenous doses of MRX-4 from 150 mg to 1800 mg
  Interventions: Drug: Single intravenous doses of MRX-4
- Single intravenous doses of placebo (Placebo Comparator): Single intravenous doses of placebo to match MRX-4
  Interventions: Drug: Single intravenous doses of placebo
- Multiple intravenous doses of MRX-4 (Active Comparator): Twice daily escalating intravenous doses of MRX-4 for 10 days: 600 mg, 900 mg, 1200 mg, and 1500 mg
  Interventions: Drug: Multiple intravenous doses of MRX-4
- Multiple intravenous doses of placebo (Placebo Comparator): Twice daily intravenous doses of placebo to match MRX-4 for 10 days
  Interventions: Drug: Multiple intravenous doses of placebo
- Single dose of intravenous and oral MRX-4 (Active Comparator): Crossover of single dose of intravenous and oral MRX-4
  Interventions: Drug: Single dose of intravenous and oral MRX-4

INTERVENTIONS:
Drug: Single intravenous doses of MRX-4 — Intravenous single escalating doses of MRX-4
  Arms: Single intravenous doses of MRX-4
Drug: Single intravenous doses of placebo — Intravenous single doses of placebo to match MRX-4
  Arms: Single intravenous doses of placebo
Drug: Multiple intravenous doses of MRX-4 — Multiple ascending doses of MRX-4 given intravenously twice daily for 10 days
  Arms: Multiple intravenous doses of MRX-4
Drug: Multiple intravenous doses of placebo — Multiple doses of placebo to match MRX-4 given intravenously twice daily for 10 days
  Arms: Multiple intravenous doses of placebo
Drug: Single dose of intravenous and oral MRX-4 — Crossover single dose of intravenous and oral MRX-4 given on Day 1 and Day 4
  Arms: Single dose of intravenous and oral MRX-4

SUMMARY:
A Phase 1 study of the safety, tolerability, and pharmacokinetics of a new oxazolidinone antibiotic. In Part 1 cohorts of healthy adults will participate in a single dose escalation study of increasing intravenous doses of MRX-4. In Part 2 cohorts of healthy adults will participate in a multiple dose escalation study of increasing intravenous doses of MRX-4 given twice daily for ten days. Part 3 is a crossover study of oral MRX-4 versus a comparable intravenous dose of MRX-4 to determine bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Underlying hepatic, renal, metabolic, hematologic, cardiovascular, or immunologic disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety of single and multiple ascending doses of MRX-4 | Screening through end of study visit on Day 7 (Part 1), Day 17 (Part II) and Day 15 (Part III)
  Summary statistics of the number of subjects with changes in vital signs, physical examinations, clinical lab data, ecg parameters, and adverse events

SECONDARY OUTCOMES:
Plasma concentration time data for MRX-4 and its metabolites | Pre-dose through 72 hours post dose
  Individual and mean plasma concentration time data for MRX-4 and its metabolites
Bioavailability of MRX-I and other MRX-4 metabolites | Pre-dose through 72 hours post dose
  Levels of MRX-4 and its metabolites in blood
Comparison of the pharmacokinetics of oral versus intravenous MRX-4 and its metabolites | Pre-dose through 72 hours post dose
  Levels of MRX-4 and its metabolites in blood
Elimination of MRX-4 and its metabolites in the urine following single dose adminstration | Pre-dose through 72 hours post dose
  Levels of MRX-4 and its metabolites in urine

IPD SHARING:
Plan to Share IPD: No